CLINICAL TRIAL: NCT03903679
Title: Is Endotracheal Tube Use Mandatory in Patients Undergoing Nasal Septum Surgery? Randomized, Controlled, Prospective Clinical Trial
Brief Title: Is Endotracheal Tube Use Mandatory in Patients Undergoing Nasal Septum Surgery?
Acronym: LMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Erol Karaaslan, Asst. Prof. Erol Karaaslan, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: erolkaraaslan2
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Airway Aspiration; Airway Complication of Anesthesia
Keywords: Airway management; Septal surgery; Laryngeal mask airway; Endotracheal tube; Presence of tracheal blood
MeSH Terms: interventions — Laryngeal Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laryngeal mask airway (Active Comparator): Patients will be maintained with laryngeal mask airway supreme during the septal surgery.
  Interventions: Device: Laryngeal mask airway
- Endotracheal tube (Sham Comparator): Patients will be maintained with endotracheal tube during the septal surgery.
  Interventions: Device: Endotracheal tube

INTERVENTIONS:
Device: Laryngeal mask airway — Patients will be maintained with laryngeal mask airway during the septal surgery.
  Arms: Laryngeal mask airway
Device: Endotracheal tube — Patients will be maintained with endotracheal tube during the septal surgery.
  Arms: Endotracheal tube

SUMMARY:
The efficacy of supraglottic airway device use in many surgeries has been shown. Due to concerns such as tracheal blood leakage and vocal cord contamination in nasal septum surgery, there are doubts about the use of laryngeal mask airway among anesthesiologists.

The primary purpose of this study is; the aim of this study was to evaluate the tracheal blood leak with a flexible fiberoptic endoscope in patients who underwent nasal septum surgery and continued airway patency via laryngeal mask airway or endotracheal tube. Secondly, oropharyngeal leak pressure, hemodynamic response, airway reflexes (laryngospasm, bronchospasm, cough, desaturation), postoperative nausea, vomiting, sore throat, hoarseness and difficulty in swallowing will be evaluated.

DETAILED DESCRIPTION:
Airway management is one of the main issue of anesthesia practice. The use of endotracheal tubes has been accepted as the standard method for many years. High pressure and long-term use of cuffed tubes related to mucosal hypoperfusion and submucosal stenosis are important. The laryngeal mask airway is produced in the 1980s and considered as a supraglottic airway used to provide airway clearance in short-term surgical procedures. The laryngeal mask airways have recently found to use in many general anesthesia applications as a minimally invasive airway method and continue to be used increasingly. More appropriate supraglottic airway vehicles with different characteristics in terms of efficacy and side effects are being developed.

Laryngeal mask airway-Supreme™ is latex-free, semi-rigid, elliptical and anatomical shape due to the fingers in the mouth of the patient easily and quickly without inserting the new generation laryngeal mask airways. Designed to provide higher sealing pressures than the laryngeal mask airway-classic. In addition, the presence of a gastric canal for gastric tube passage is another important advantage.

The efficacy of supraglottic airway device use in many surgeries has been shown. Due to concerns such as tracheal blood leakage and vocal cord contamination in nasal septum surgery, there are doubts about the use of laryngeal mask airway among anesthesiologists.

The primary purpose of this study is; the aim of this study was to evaluate the tracheal blood leak with a flexible fiberoptic endoscope in patients who underwent nasal septum surgery and continued airway patency via laryngeal mask airway or endotracheal tube. Secondly, oropharyngeal leak pressure, hemodynamic response, airway reflexes (laryngospasm, bronchospasm, cough, desaturation), postoperative nausea, vomiting, sore throat, hoarseness and difficulty in swallowing will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old,
* American Society of Anesthesiologists I-II
* Patients with elective nasal septum surgery.
* Patients who agreed to participate with informed consent form.

Exclusion Criteria:

* Under 18 years,
* Over 65 years,
* American Society of Anesthesiologists III-IV,
* Patients with severe respiratory, hepatic or renal dysfunction,
* Patients with history of allergy to anesthesia medications
* Modified mallampati grade 4,
* Thyromental distance <65 mm,

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-04-05 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-08 (Actual)

PRIMARY OUTCOMES:
Presence of blood in trachea | From the time 2minutes after the septal surgery to the time of extubation
  Presence of blood in trachea will be evaluated on a scale and it is defined as the level of presence of blood on glottis-trachea and distal trachea. (1 = no, 2 = mild, 3 = moderate, 4 = severe).

SECONDARY OUTCOMES:
Sore-throat | From the time 10 minutes after awakening from anesthesia to the time 24 hours postoperatively
  Sore-throat is defined as constant pain felt independently of swallowing. The evaluation was made with 0 ile10 numerical pain rating scale. According to numerical pain rating scale, sore throat score was evaluated as; 0-1 none, 2-4 between mild, 5-7 intermediate and 8-10 severe N
Oropharyngeal leak pressure | From the time 2 minutes after anesthesia induction to the correction of inserted device 5 minutes after anesthesia induction
  Oropharyngeal leak pressures were measured while the head was in neutral position. The flowmeter oxygen current was set at 3 L/min and the expiratory valve was closed. When an investigator who did not know which type of airway device was placed, another researcher looked at the current pressure value from the aneroid manometer and confirmed that the pressure remained constant (pressure gauge stability test). This value was recorded as the value of Oropharyngeal leakage pressure. To prevent lung exposure to barotrauma, the expiratory valve was opened when the peak inspiratory pressure reached 40 pressure, and the test was terminated.

CONTACTS AND LOCATIONS:
Overall Officials: Erol Karaaslan, Asst. Prof., Principal Investigator — Inonu University Medical Faculty
Locations (1):
- Inonu University Medical Faculty, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mao S, Du X, Ma J, Zhang G, Cui J. A comparison between laryngeal mask airway and endotracheal intubation for anaesthesia in adult patients undergoing NUSS procedure. J Thorac Dis. 2018 Jun;10(6):3216-3224. doi: 10.21037/jtd.2018.05.74. PMID 30069317
- [Derived] Karaaslan E, Akbas S, Ozkan AS, Colak C, Begec Z. A comparison of laryngeal mask airway-supreme and endotracheal tube use with respect to airway protection in patients undergoing septoplasty: a randomized, single-blind, controlled clinical trial. BMC Anesthesiol. 2021 Jan 7;21(1):5. doi: 10.1186/s12871-020-01222-4. PMID 33407130

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-28): https://cdn.clinicaltrials.gov/large-docs/79/NCT03903679/Prot_SAP_000.pdf